CLINICAL TRIAL: NCT02290990
Title: A Randomized Controlled Trial on Integrated Imaginative Distention in MS Ans Insomnia: a Self Managed Tool to Cope With Fatigue, Stress and Insomnia
Brief Title: Efficacy Study of "Imaginative Distention", a Self Managed Tool to Cope With Fatigue,Insomnia and Stress in pw Insomnia and pw MS
Acronym: DIMMISI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIMMI SI
Record Dates: First submitted 2014-10-07; First posted 2014-11-14 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Multiple Sclerosis patients (Experimental): Patients with MS
  Interventions: Behavioral: "Imaginative Distention" technique
- Insomnia patients (Experimental): Patients with insomnia
  Interventions: Behavioral: "Imaginative Distention" technique
- Health professionists (Experimental): Health professionists as healthy volunteers
  Interventions: Behavioral: "Imaginative Distention" technique
- Waiting list MS (Active Comparator): pw MS filled the self administered questionnaire but they receive any training. They must wait study conclusion to be treated
  Interventions: Behavioral: "Imaginative Distention" technique
- Waiting list arm Insomnia (Active Comparator): pw INS Insomnia Subject filled the self administered questionnaire but they receive any training. They must wait study conclusion to be treated
  Interventions: Behavioral: "Imaginative Distention" technique
- Waiting list arm Health professionists (Active Comparator): Health professionist filled the self administered questionnaire but they receive any training. They must wait study conclusion to be treated.
  Interventions: Behavioral: "Imaginative Distention" technique

INTERVENTIONS:
Behavioral: "Imaginative Distention" technique — ID is an Imaginative relaxation technique which combines physical and mental relaxation. ID technique reaches physical relaxation through planned alternated movements taken from Jacobson PMRT which consist of specific muscle contractions and subsequent relaxations, with a precise temporal scanning. Psychological relaxation is achieved thanks to mental imagery (motor imagery, body scan, imagination).

SUMMARY:
Imaginative Distention (ID) is proposed as supportive and integrative intervention to cope with fatigue, (principal end point), to cope with insomnia, stress perception and to improve QoL of pw MS, insomnia pw and health care personnel. ID is safe and it can be easily learned and practised without of any particular instrument and also feasible in disabled pw. This technique allows persons to experience the body as a source of well-being and not just fatigue, pain and disease. ID can become a self managed tool of empowerment to cope with MS, to reduce its negative impact on daily life and job performances. Adherence to pharmacological therapies could be improved using ID.

For pw MS ID could have specific and customizable rehabilitation implications to improve motor disability, as already seen in stroke patients. The principal end point of the trial is verify ID efficacy on fatigue and its specificity on pw MS at the end of the training. For this reason, ID efficacy will be tested in comparative terms too. Among all possible comparison populations, we selected: pw insomnia, which is stress related disease and health personnel, because at risk of stress. The control groups comparison permits to evaluate the specificity of ID on pw MS. The three groups are randomised to intervention or waiting list. The training is 8 weekly session long. Self administered questionnaire are filled by participants before and after the training, and 3-6 months later. The extent of change in outcome measure monitored in each exposed group vs. unexposed will allow to separate the non-disease specific effect of ID from the MS-specific effect. The difference in estimates will allow to determine the extent of the true effect of ID in pw MS. All outcome measure will be compared among all groups mentioned and over time. The study would identify also the most important outcome measures for MS patients questioning them in a focus group. This aspect is very important because could differs from which clinicians and researchers think about.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic neurological disorder with physical, emotional and cognitive symptoms. The diagnosis and the unpredictable and variable nature of the disease have profound social and psychological impact on persons with MS (pw MS). Fatigue, depression and disability are independent determinants of quality of life (QoL) and it is known that different kinds of stress may impact on disease activity. The "Imaginative Distention" (ID) is a mind-body technique that combines relaxation, imagination and motor imagery. ID derives from Progressive Muscle Relaxation Technique (PMRT) that was shown effective on fatigue in MS and in cancer patients, as well as cognitive behavioural psychotherapy, which includes relaxation. Mind-body modalities appear safe. ID can be easily learned and practised without any particular instrument and is also feasible in disabled pw MS. The aim of our study is to evaluate the effectiveness of ID as supportive and integrative intervention to cope with MS. We plan the first randomized controlled study (RCT) that will investigate the effectiveness of ID on fatigue (primary end point), disease specific QoL, insomnia, stress perception and physiological parameters. The primary outcome is the change in fatigue recorded post-intervention. Fatigue has a generically stress-related and a specifically disease-related component. To estimate the effect of ID on the specific MS-related component of fatigue, we will also monitor two additional groups of subjects, one with insomnia (with fatigue and poor QoL but with lesser impact on health condition) and one under generic stress (health professionals, with fatigue and normal to poor QoL and limited if any impact on health condition). Each study group - MS, insomnia, health professionals - will be randomised 1:1 to intervention or waiting list. The design is therefore parallel, randomised, controlled vs. no intervention, open, stratified by condition. Enrolment is voluntary. All participants will undergo a pre-evaluation visit which includes four self administered questionnaires (MFIS for fatigue, VRS Verbal Rating Scale for stress, ISI Insomnia Severity Index, MSQOL-54 Multiple Sclerosis Quality of Life), the EDSS Expanded Disability Status Scale and a brief cognitive screening for pw MS. After randomization, ID is practiced in groups, once a week, for two months. At the end, pw MS will be involved in focus groups to identify the agreement between investigator selected and patients-expected relevance of the outcomes used in the study, as well as other outcomes of relevance for the patients but not monitored in the study, to be possibly implemented in future trials. Follow up evaluations at two, five and eight months will include EDSS and the self-administered questionnaires and, at five months, the cognitive screening. If efficacy will be proved, ID could become a tool of empowerment to cope with MS, to reduce its negative impact on daily life and job performances and, possibly, to improve the adherence to pharmacological therapies.

ELIGIBILITY:
Inclusion Criteria:

* any gender, ethnicity
* aged 18-65 years
* ability to understand Italian to be able to conduct the study
* adherence to the study by written informed consent
* absence of serious internal medicine and psychiatric comorbidities

Exclusion Criteria:

* under 18 and above 65 years
* lack of understanding Italian to conduct of the studies
* inability to provide informed consent
* presence of severe internal medicine and psychiatric comorbidities

Specific criteria for inclusion:

Pw MS:

* Diagnosis according to the criteria of Polman, 2011: relapsing remitting or progressive (primary and secondary)
* Or in no specific drug therapy for the disease and symptomatic

Pw insomnia:

* Diagnosis of psychophysiological insomnia according to DSM IV
* Or in no specific drug therapy for the disease and symptomatic

Healthy professionals:

- Healthy personnel operating within the Niguarda Hospital

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Fatigue | Change from baseline in MFIS score at two months + one week
  Evaluated with MFIS self administered questionnaire.Modified Fatigue Impact Scale (MFIS) is a self-assessment,values fatigue on daily life impact. Provides 21 items with 5-point Likert scale answer (from 0 = never to 4 = almost always).Total score ranges from 0 to 84 and includes three subscales:physical,cognitive and psychosocial fatigue (score ranges between 0-8)

SECONDARY OUTCOMES:
Quality of life | month 2;month 3;month 6
  Includes 54 items which generate 12 subscales with two summary scores, and two additional measures given by the single item.
Stress | month 2;follow-up (month 3;month 6)
  It consists of 15 items and breaks down into five areas of evaluation which, when added, quantify the stress response: anxiety, depression, somatization, aggression, social support
Insomnia | month 2
  Consists of 7 items answered on a 4-point Likert scales, refers to the Mental Disorders Manual DSM-IV criteria for insomnia, and assesses the Individual impact of the symptoms in the last 2 weeks
Physiological parameters and Neurological evaluation | month 2,month 3;month 6
  The EDSS is the most widely used to assess neurological disability with a score between 0 and 10
Cognitive screening | baseline,month 3
  Symbol Digit Modalities Test. Points 0-120. The California Verbal Learning Test - Second Edition. Points: 0-16 Visuospatial Memory Test - Revised. It takes 15 minutes. Points 0-36

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ospedaliera Ospedale Niguarda Ca' Granda, Milan, Italy

REFERENCES:
- [Derived] Sgoifo A, Bignamini A, La Mantia L, Celani MG, Parietti P, Ceriani MA, Marazzi MR, Proserpio P, Nobili L, Protti A, Agostoni EC. Integrated Imaginative Distention Therapy to Cope with Fatigue. DIMMI SI Study: The First Randomized Controlled Trial in Multiple Sclerosis. Neurol Ther. 2017 Dec;6(2):213-223. doi: 10.1007/s40120-017-0081-9. Epub 2017 Aug 9. PMID 28795383